CLINICAL TRIAL: NCT01066234
Title: A Randomized Phase II Study of Adjuvant Concurrent Chemoradiotherapy vs Chemotherapy Alone in Completely Resected Microscopic N2 Non-small Cell Lung Cancer
Brief Title: Adjuvant CCRT vs CT in Minimal N2 NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Keunchil Park, Principal investigator, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-04-004
Record Dates: First submitted 2010-02-08; First posted 2010-02-10 (Estimated); Last update posted 2021-03-22 (Actual); Status verified 2021-03

CONDITIONS: Non-small Cell Lung Cancer
Keywords: Microscopic N2 Non-small Cell Lung Cancer; Paclitaxel; Carboplatin; Cisplatin
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Chemoradiotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- concurrent chemoradiotherapy (Experimental)
  Interventions: Radiation: concurrent chemoradiotherapy
- chemotherapy only (Active Comparator)
  Interventions: Drug: chemotherapy only

INTERVENTIONS:
Radiation: concurrent chemoradiotherapy — weekly paclitaxel 50mg/m2 plus weekly cisplatin 25mg/m2 5times with concurrent radiotherapy (5000rad/25fx) for 5 weeks followed by 2 cycles of 3-weekly paclitaxel (175mg/m2) plus cisplatin 80mg/m2.
  Arms: concurrent chemoradiotherapy
Drug: chemotherapy only — four cycles of 3-weekly paclitaxel (175mg/m2) and carboplatin (AUC5.5).
  Arms: chemotherapy only

SUMMARY:
This study propose adjuvant concurrent chemoradiotherapy vs chemotherapy alone in completely resected microscopic N2 NSCLC

DETAILED DESCRIPTION:
Approximately 15% of patients with non-small cell lung cancer are diagnosed with stage IIIA-N2 disease. However, this subgroup is heterogeneous, with lymph nodes that are only microscopically invaded to those that are radiologically visible with bulky ipsilateral mediastinal lymph node involvement. Surgical resection in selected patients results in 5-year survival rates of 7-24%.

The standard treatment for locally advanced clinical N2 disease is definitive concurrent chemoradiotherapy or induction chemotherapy (± radiation) followed by operation. However, in some patients, N2 status could be confirmed only after curative operation without any evidence of N2 diseases through preoperative evaluation methods (CT, PET, mediastinoscopy). We usually define those N2 disease found only after curative operation as microscopic N2, and do adjuvant chemotherapy, radiotherapy or concurrent chemoradiotherapy. However, little data about the adjuvant therapy for completely resected N2 disease have been available, Hence, we propose a randomized phase II study of adjuvant concurrent chemoradiotherapy vs chemotherapy alone in completely resected microscopic N2 NSCLC.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of stage IIIA(N2) NSCLC that was completely resected by lobectomy, bilobectomy, pneumonectomy, or sleeve lobectomy through any incision (thoracoscopic or video-assisted thorascopic surgery approaches were acceptable)
2. "Pathologic N2" disease (involvement of N2 nodes can only be determined at the time of surgical exploration or postoperative pathologic analysis)
3. Age ≥18years
4. No known residual disease (negative resection margin and no extracapsular invasion of lymph node metastasis)
5. ECOG performance status of 0 to 1
6. No previous chemotherapy or RT
7. Adequate organ function as evidenced by the following; Absolute neutrophil count > 1.5 x 109/L; platelets > 100 x 109/L; total bilirubin ≤1.5 UNL; AST and/or ALT < 5 UNL; creatinine clearance ≥ 50mL/min
8. Written informed consent form

Exclusion Criteria:

1. Patients with preoperative mediastinoscopic N2 positive disease
2. Uncontrolled systemic illness such as DM, CHF, unstable angina, hypertension or arrhythmia
3. Patients with post-obstructive pneumonia or uncontrolled serious infection
4. Pregnant or nursing women ( Women of reproductive potential have to agree to use an effective contraceptive method)
5. Prior history of malignancy within 5 years from study entry except for a adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer, well-treated thyroid cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2021-01-18 (Actual); Study Completion 2021-01-18 (Actual)

PRIMARY OUTCOMES:
Disease-free survival | 36 months

SECONDARY OUTCOMES:
Overall survival (OS) | 36 months
Pattern of relapse | 36 months
Toxicity profile | 36 months
Quality of life (QOL) | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Keunchil Park, M.D., Ph.D, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Sun JM, Noh JM, Oh D, Kim HK, Lee SH, Choi YS, Pyo H, Ahn JS, Jung SH, Ahn YC, Kim J, Ahn MJ, Zo JI, Shim YM, Park K. Randomized Phase II Trial Comparing Chemoradiotherapy with Chemotherapy for Completely Resected Unsuspected N2-Positive Non-Small Cell Lung Cancer. J Thorac Oncol. 2017 Dec;12(12):1806-1813. doi: 10.1016/j.jtho.2017.09.1954. Epub 2017 Sep 28. PMID 28962948